CLINICAL TRIAL: NCT06548750
Title: Intrinsic vs Combined Foot Muscle Strengthening for Pes Planovalgus in Preschoolers: A Randomized Controlled Trial
Brief Title: Foot Muscle Strengthening Exercises for Pes Planovalgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DT2024-AE
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pes Planus
Keywords: Intrinsic foot muscle; Physiotherapy; Foot core; Flat foot; Extinsic foot muscle
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Intervention Model Description: There will be an equal number of participants in the two groups randomized by the computer
Who Masked: Investigator
Masking Description: The assessor will not know which participant received which intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Individuals with a diagnosis of pes planovalgus who underwent supervised exercise under the guidance of a physiotherapist for 8 weeks, 1 day a week.
  Interventions: Other: Intrinsic and Ectrinsic Exercise
- Control Group (Active Comparator): Individuals with a diagnosis of pes planovalgus who underwent supervised exercise under the guidance of a physiotherapist for 8 weeks, 1 day a week.
  Interventions: Other: Intrinsic Exercise

INTERVENTIONS:
Other: Intrinsic and Ectrinsic Exercise — Intrinsic and extrinsic muscle strengthening exercises
  Arms: Intervention Group
Other: Intrinsic Exercise — Intrinsic muscle strengthening exercises
  Arms: Control Group

SUMMARY:
Pes planovalgus is a common foot condition affecting the child population. It is characterized by the partial or complete collapse of the medial longitudinal arch with rearfoot eversion and forefoot abduction, which is associated with changes in lower extremity kinematics during dynamic activity.

The lower extremity chain includes the foot, ankle, knee, and hip joints, with the feet acting as the base of support. However, due to their small size, maintaining balance can be challenging. Any small dynamic change in the foot, as the support base, can impact overall body posture. The foot arch, which can be pronated or supinated, affects proprioceptive input by altering joint movement, contact area, and muscle strategy for stability. Pes planovalgus, characterized by excessive subtalar pronation, lead to instability and hypermobility, requiring more neuromuscular control to maintain balance. As a result, flat feet can cause pathomechanical issues and compensatory actions in the lower extremity chain, affecting overall body balance.

The effectiveness of exercise interventions, particularly foot intrinsic muscle strengthening exercises, in increasing the medial longitudinal arch in individuals with pes planus has been investigated in numerous studies. It is widely accepted that both intrinsic and extrinsic muscle groups play a crucial role in the formation, maintenance, and enhancement of foot arches. However, there is a lack of studies specifically examining the effectiveness of exercises aimed at strengthening these muscles in children with pes planovalgus. Therefore, the purpose of this study is to compare the effects of two corrective exercise programs focused on the improvement of the medial longitudinal arch in children with pes planovalgus: one incorporating routine intrinsic muscle exercises and the other combining them with extrinsic muscle exercises.

DETAILED DESCRIPTION:
Voluntary children who have been diagnosed with pes planovalgus will be included in the study. Signed voluntary consent will be obtained from caregivers. Participants will be divided into two groups. Study groups will be as follows: a) Intervention Group (Intrinsic&Extrinsic Exercise), b) Control Group (Intrinsic Exercise).

ELIGIBILITY:
Inclusion Criteria:

* Presence of bilateral pes planovalgus,
* Being between 4-7 years of age,
* Having a body mass index within normal limits

Exclusion Criteria:

* Having high femoral anteversion, internal tibial torsion and metatarsus adductus
* Having leg length inequality
* Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
* Having a history of pain, deformity or surgery related to the vertebral column and lower extremities
* Having a cognitive, mental or serious psychiatric disease
* Having been involved in any exercise program or sports activity in the last six months

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
Single Leg Stance Test | change from baseline balance at 2 months
  It evaluates the participants' standing balance. The entire lower extremity will be positioned in full extension, while the other side will be positioned in 90 degree flexion of the lower extremity hip and knee. The time will be started when the participants' eyes are closed and the untested feet lose contact with the ground, and the time will be stopped when they put their feet back on the ground or when their body sway increases too much.
Timed-up and Go Test | change from baseline balance at 2 months
  TUG is a measure of dynamic balance and the risk of falling. It entails individuals rising from a chair, walking a distance of 3 feet, turning, and then sitting back down.

SECONDARY OUTCOMES:
Range of Motion | 2 times for 8 weeks
  For goniometric measurement, the pivot point will be placed on the lateral malleolus. The fixed arm will be held parallel to the lateral midline of the fibula. The mobile arm will follow the lateral midline of the 5th metatarsal bone.
Thomas Test | 2 times for 8 weeks
  The Thomas Test will be used to determine the shortness of the hip flexors. The Thomas test is performed with the patient in the supine position with the gluteal folds on the short side of the stretcher. The untested side lower extremity is pulled towards the abdomen by performing hip-knee flexion; the tested side extremity is checked to see if it is separated from the stretcher.
Duncan-Ely Test | 2 times for 8 weeks
  The Duncan-Ely test will be used to assess rectus femoris spasticity and shortness. In this test, the patient will be asked to lie in a prone position. The physiotherapist will attempt to quickly and passively bring the patient's knee joint on the side being assessed into full flexion. If the heel cannot touch the hip or the hip on the side being tested lifts off the stretcher, the test is considered positive.
Popliteal Angle Assessment | 2 times for 8 weeks
  It will be used to detect hamstring shortness. The patient will be in the supine position, the tested side hip-knee will be flexed to 90°, and then passive extension will be applied to the knee. Goniometric measurement will be made when the end-feel is felt in the patient's knee joint.
Navicular Drop Test (NDT) | 2 times for 8 weeks
  It is one of the static foot assessment tools and represents the sagittal plane displacement of the navicular tuberosity in a neutral position. If the NDT is below 5 mm, the foot is in supination; if it is between 6-8 mm, the foot is neutral; and if it is above 9 mm, the foot is in pronation.
Foot Posture Index-6 (FPI-6) | 2 times for 8 weeks
  FPI-6, which is a simple, fast and reliable method applicable to pediatric feet, defines the static postural analysis of the foot when equal load is applied to both feet during standing. Scores of 0-5 define normal foot; 6-9 define pes planovalgus and 10-12 define advanced pes planovalgus.
6-minutes Walking Test | 2 times for 8 weeks
  It is a useful test to assess functional exercise capacity. Patients are asked to walk as fast as they can down a straight 30-meter corridor for six minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Tuncer, PhD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Huang C, Chen LY, Liao YH, Masodsai K, Lin YY. Effects of the Short-Foot Exercise on Foot Alignment and Muscle Hypertrophy in Flatfoot Individuals: A Meta-Analysis. Int J Environ Res Public Health. 2022 Sep 22;19(19):11994. doi: 10.3390/ijerph191911994. PMID 36231295
- [Background] Hara S, Kitano M, Kudo S. The effects of short foot exercises to treat flat foot deformity: A systematic review. J Back Musculoskelet Rehabil. 2023;36(1):21-33. doi: 10.3233/BMR-210374. PMID 35871320
- [Background] Okamura K, Fukuda K, Oki S, Ono T, Tanaka S, Kanai S. Effects of plantar intrinsic foot muscle strengthening exercise on static and dynamic foot kinematics: A pilot randomized controlled single-blind trial in individuals with pes planus. Gait Posture. 2020 Jan;75:40-45. doi: 10.1016/j.gaitpost.2019.09.030. Epub 2019 Sep 29. PMID 31590069
- [Background] Pabon-Carrasco M, Castro-Mendez A, Vilar-Palomo S, Jimenez-Cebrian AM, Garcia-Paya I, Palomo-Toucedo IC. Randomized Clinical Trial: The Effect of Exercise of the Intrinsic Muscle on Foot Pronation. Int J Environ Res Public Health. 2020 Jul 7;17(13):4882. doi: 10.3390/ijerph17134882. PMID 32645830
- [Background] Haun C, Brown CN, Hannigan K, Johnson ST. The Effects of the Short Foot Exercise on Navicular Drop: A Critically Appraised Topic. J Sport Rehabil. 2020 May 8;30(1):152-157. doi: 10.1123/jsr.2019-0437. PMID 32384261
- [Background] Moon DC, Kim K, Lee SK. Immediate Effect of Short-foot Exercise on Dynamic Balance of Subjects with Excessively Pronated Feet. J Phys Ther Sci. 2014 Jan;26(1):117-9. doi: 10.1589/jpts.26.117. Epub 2014 Feb 6. PMID 24567688
- [Derived] Tuncer D, Erekdag A, Senaran H, Uzer G. Intrinsic vs. combined foot muscle strengthening for pes planovalgus in children aged 4-7 years: a randomized controlled trial. Eur J Pediatr. 2025 Sep 25;184(10):636. doi: 10.1007/s00431-025-06480-3. PMID 40999032